CLINICAL TRIAL: NCT03988374
Title: Clinical Efficacy Evaluation of Three Dentifrices Containing 35%, 20%, and 0% Sodium Bicarbonate on the Reduction of Plaque and Gingivitis
Brief Title: Clinical Efficacy Evaluation of Three Dentifrices
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ST-7700
Record Dates: First submitted 2019-04-04; First posted 2019-06-17 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-04

CONDITIONS: Gingival Inflammation and Bleeding; Dental Plaque
MeSH Terms: conditions — Gingivitis; Hemorrhage; Dental Plaque | interventions — Dentifrices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 0% Baking Soda Dentifrice (Active Comparator)
  Interventions: Drug: Dentifrices
- 20% Baking Soda Dentifrice (Active Comparator)
  Interventions: Drug: Dentifrices
- 35% Baking Soda Dentifrice (Active Comparator)
  Interventions: Drug: Dentifrices

INTERVENTIONS:
Drug: Dentifrices — Dentifrice on plaque, gingivitis, and bleeding.

SUMMARY:
Clinical study to evaluate and compare the efficacy of two baking soda containing dentifrices, containing 20% and 35% baking soda, to a non-baking soda dentifrice for their ability to reduce gingivitis and plaque following 6-months of use.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent prior to being entered into the study.
* Be between 18 and 70 years of age, male or female.
* Have at least eighteen (18) natural teeth with scorable facial and lingual surfaces as determined by the Examiner. Teeth that are grossly carious, orthodontically banded, exhibiting general cervical abrasion and/or enamel abrasion, or third molars will not be included in the tooth count.
* Have a mean baseline plaque index score ≥ 1.95 as determined by the Soparkar Modification of the Turesky Modification of the Quigley-Hein Plaque Index (Pl).
* Have a mean baseline gingival index score of ≥ l.70 and ≤ 3.0 as determined by the Modified Gingival Index (MGI).
* Presence of ≥ 10 bleeding sites upon probing.
* Agree not to have a dental prophylaxis or any other elective, non-emergency dental procedures any time during the study.
* Agree to abstain from the use of chewing gum, mouth rinses, any toothpaste other than the study toothpaste, tooth whitening products (either professional or at home use) and all other oral hygiene other than the study procedures for the duration of the study.
* Agree to refrain from all oral hygiene on the morning of each evaluation visit and to refrain from eating, drinking, and smoking for 4 hrs, prior to each evaluation visit.
* Agree to comply with the conditions and schedule of the study.

Exclusion Criteria:

* Physical limitations or restrictions that might preclude normal tooth brushing.
* Evidence of gross oral pathology, including widespread caries or chronic neglect, extensive restoration, preexisting gross plaque or soft or hard tissue tumor of the oral cavity.
* Heavy supra- or subgingival calculus that might interfere with evaluations as determined by the Investigator/Examiner.
* Evidence of major oral hard or soft tissue lesions or trauma at the baseline visit as determined by the Investigator/Examiner.
* Conditions requiring antibiotic treatment prior to dental procedures.
* History of uncontrolled diabetes or hepatic or renal disease, or other serious conditions or transmittable diseases, (e.g. cardiovascular disease, AIDS).
* Subjects with grossly carious, fully crowned, or extensively restored teeth, orthodontic appliances, peri/oral piercings, or removable partial dentures.
* Treatment with antibiotics within the 1-month period before the baseline examination, or a condition that is likely to require antibiotic treatment over the course of the trial.
* Chronic treatment (2 weeks or more) with any medication known to affect periodontal status (including phenytoin, calcium antagonists, cyclosporine, coumarin, nonsteroidal anti-inflammatory drugs, and aspirin) within 1 month of the baseline examination. All other medications for chronic medical conditions must have been initiated at least 3 months before enrollment.
* Have severe periodontal disease or being actively treated for periodontal disease.
* Having history of early-onset periodontitis or acute necrotizing ulcerative gingivitis.
* Concomitant periodontal therapy other than prophylaxis in the last 6 months.
* Professional prophylaxis within 1 month prior to the baseline clinical evaluation.
* Subjects who participated in a gingivitis study in the past month.
* Daily use of chemotherapeutic antiplaque/antigingivitis products within the past 4 months.
* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses.
* Subjects who are allergic to any ingredients in the test or control product, as listed on the IRB Safety Assessment.
* Self-reported pregnancy and nursing since hormonal changes can exaggerate gingival response to dental plaque.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- All Sum Research Center Ltd., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 0% Baking Soda Dentifrice: Dentifrice, not containing baking soda, evaluated for ability to reduce gingivitis and plaque following 6-months of use.
- 20% Baking Soda Dentifrice: Dentifrice, containing 20% baking soda, evaluated for ability to reduce gingivitis and plaque following 6-months of use.
- 35% Baking Soda Dentifrice: Dentifrice, containing 35% baking soda, evaluated for ability to reduce gingivitis and plaque following 6-months of use.
Period: Overall Study
Arm/Group | 0% Baking Soda Dentifrice | 20% Baking Soda Dentifrice | 35% Baking Soda Dentifrice
Started | 104 | 107 | 108
Completed | 103 | 105 | 107
Not Completed | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0% Baking Soda Dentifrice | 20% Baking Soda Dentifrice | 35% Baking Soda Dentifrice | Total
Number analyzed (Participants) | 103 | 105 | 107 | 315
Age, Continuous [Mean (Full Range); unit: Age] | 44.07 [18 to 70] | 47.50 [18 to 70] | 47.32 [18 to 70] | 46.3 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 80 | 229
  Male | 28 | 31 | 27 | 86
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 103 | 105 | 107 | 315
Gingvial Efficacy [Mean (Full Range); unit: units on a scale] — Measure Description: Lobene Modified Loe-Silness Gingival Scoring Index (MGI) - gingival sites were visually scored at each visit on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth, using a scale of 0-4. Lower values represent a better outcome.
  units on a scale | 2.081 [0 to 4] | 2.094 [0 to 4] | 2.092 [0 to 4] | 2.089 [0 to 4]
Gingival Bleeding Efficacy [Mean (Full Range); unit: units on a scale] — Measure Description: Bleeding was assessed on all scorable buccal and lingual surfaces by inserting a periodontal probe into the gingival crevice and sweeping from the distal aspect to the mesial aspect around the tooth at a depth of approximately 1 mm and angle of approximately 60 degrees while in contact with the sulcular epithelium. Three areas (distobuccal, midbuccal and midlingual) were assessed around each tooth. Sites were scored at each visit using the Gingival Bleeding Index (GBI) as defined by Saxton and van der Ouderaa on a scale of 0-2. Lower values represent a better outcome.
  units on a scale | 0.165 [0 to 2] | 0.178 [0 to 2] | 0.189 [0 to 2] | 0.177 [0 to 2]
Plaque Efficacy [Mean (Full Range); unit: units on a scale] — Measure Description: Plaque was scored at each visit using the Soparker modification of the Turesky Modification of the Quigley-Hein Plaque Index (PI) on all scorable buccal and lingual surfaces. Plaque was stained with disclosant and each tooth was divided into six areas for scoring on a scale of 0-5. A PI score for each subject was calculated by adding all individual site scores (6 per tooth) and dividing by the total number of sites scored (teeth x 6). Lower values represent a better outcome.
  units on a scale | 2.409 [0 to 5] | 2.411 [0 to 5] | 2.356 [0 to 5] | 2.4 [0 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Mean Within-Treatment Whole-Mouth Score - Gingival Efficacy
Description: Mean Within-Treatment Whole-Mouth Score as measured by Gingival Index (0=absence of inflammation, 1=mild inflammation: slight change in color, little change in texture of any portion of but not the entire marginal or papillary gingival unit, 2=mild inflammation: slight change in color, little change in texture to entire marginal or papillary gingival unit, 3=moderate inflammation: glazing, redness, edema and/or hypertrophy of the marginal or papillary gingival unit, 4=severe inflammation: marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. The scale ranges from 0-4.
Time Frame: baseline, six weeks, 3 months and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0% Baking Soda Dentifrice | 20% Baking Soda Dentifrice | 35% Baking Soda Dentifrice
Number analyzed (Participants) | 103 | 105 | 107
units on a scale
  Baseline | 2.081 (0.096) | 2.094 (0.117) | 2.092 (0.106)
  6 weeks | 1.996 (0.138) | 1.919 (0.171) | 1.882 (0.174)
  3 months | 1.980 (0.155) | 1.841 (0.198) | 1.766 (0.229)
  6 months | 1.946 (0.149) | 1.763 (0.209) | 1.653 (0.256)

2. Primary Outcome: Mean Within-Treatment Whole-Mouth Score - Gingival Bleeding Efficacy
Description: Mean Within-Treatment Whole-Mouth Score as measured by Gingival Bleeding Index (0=absence of bleeding after 30 seconds, 1= bleeding observed after 30 seconds, 2= bleeding occurs instantly). The scale ranges from 0-2.
Time Frame: baseline, six week, three months, and six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0% Baking Soda Dentifrice | 20% Baking Soda Dentifrice | 35% Baking Soda Dentifrice
Number analyzed (Participants) | 103 | 105 | 107
units on a scale
  Baseline | 0.165 (0.085) | 0.178 (0.129) | 0.189 (0.114)
  6 weeks | 0.149 (0.091) | 0.135 (0.122) | 0.122 (0.081)
  3 months | 0.141 (0.088) | 0.116 (0.117) | 0.094 (0.067)
  6 months | 0.129 (0.082) | 0.096 (0.104) | 0.069 (0.053)

3. Primary Outcome: Mean Within-Treatment Whole-Mouth Score - Plaque Efficacy
Description: Mean Within-Treatment Whole-Mouth Score as measured by Plaque Index (0=no visible plaque, 1=separate flecks of plaque at the cervical margin of the tooth, 2=a thin, continuous band of plaque (up to 1mm wide) at the cervical margin, 3= a band of plaque wider than 1 mm but covering less than one-third of the crown, 4=plaque covering at least one-third but less than two-thirds of the crown, 5= plaque covering two-thirds or more of the crown). The scale ranges from 0-5.
Time Frame: baseline, six weeks, three months, and six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0% Baking Soda Dentifrice | 20% Baking Soda Dentifrice | 35% Baking Soda Dentifrice
Number analyzed (Participants) | 103 | 105 | 107
units on a scale
  Baseline | 2.409 (0.220) | 2.411 (0.244) | 2.356 (0.240)
  6 weeks | 2.280 (0.211) | 2.134 (0.259) | 2.026 (0.227)
  3 months 3 months | 2.251 (0.202) | 2.066 (0.260) | 1.907 (0.265)
  6 months | 2.196 (0.191) | 1.925 (0.239) | 1.793 (0.287)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 0% Baking Soda Dentifrice | 20% Baking Soda Dentifrice | 35% Baking Soda Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/105 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/105 | 0/107
Other Adverse Events (participants affected / at risk) | 4/103 | 17/105 | 2/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0% Baking Soda Dentifrice (N=103) | 20% Baking Soda Dentifrice (N=105) | 35% Baking Soda Dentifrice (N=107)
Primary discomforts (General disorders) | 1 (1) | 11 (11) | 0 (0) — Mild oral mucosal sloughing
Primary discomforts (General disorders) | 3 (3) | 1 (1) | 0 (0) — Mild Dry Mouth
Primary discomforts (General disorders) | 0 (0) | 2 (2) | 0 (0) — Mild oral tingling/burning sensation
Primary discomforts (General disorders) | 0 (0) | 3 (3) | 2 (2) — Mild sensitive/irritated gums/teeth

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Master service agreement and confidentiality agreement in place

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03988374/Prot_SAP_000.pdf